CLINICAL TRIAL: NCT04509011
Title: Randomized Controlled Trial of Fluobeam® LX Compared With Clinical Assessment of Parathyroid Glands to Counteract Postoperatively Failing Parathyroid Function With Low Blood Calcium After Thyroid Surgery
Brief Title: Autofluorescence vs Clinical Assessment of Parathyroid Glands During Thyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Haukeland University Hospital (Other); Jagiellonian University (Other); Sahlgrenska University Hospital (Other); Hospital Rudolfstiftung (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-05948
Record Dates: First submitted 2020-08-04; First posted 2020-08-11 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Hypoparathyroidism Postprocedural
Keywords: Hypoparathyroidism; PTH; Hypocalcemia
MeSH Terms: conditions — Hypoparathyroidism; Hypocalcemia

STUDY DESIGN:
Intervention Model Description: Intervention group (intraoperative use of Fluobeam®-LX during thyroid surgery) Control group (clinical assessment and identification of parathyroid glands during thyroid surgery)
Who Masked: Participant
Masking Description: The participant is not informed of the assigned group, whereas the the care giver (surgeon) is informed due to the use (or not) of the Fluobeam®-LX.
  Randomization is performed 1: 1 in blocks of 10 via the Eurocrine quality register platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluobeam® LX (Experimental): Fluobeam® LX is used to detect autofluorescens and identify and evaluate parathyroid glands
  Interventions: Device: Fluobeam® LX
- Control (No Intervention): In the control group, the parathyroid glands are identified and evaluated by eye (ocular examination).

INTERVENTIONS:
Device: Fluobeam® LX — Fluobeam®-LX is used to identify and evaluate parathyroid glands using auto-fluorescence during thyroid surgery.
  Arms: Fluobeam® LX

SUMMARY:
The purpose of the investigation is to study if the use of Fluobeam®-LX to identify parathyroid glands through autofluorescence during thyroid surgery, may reduce the risk of postoperative hypoparathyroidism, defined as low PTH in patients undergoing total thyroidectomy

DETAILED DESCRIPTION:
Temporary and permanent hypoparathyroidism is probably the most important complication of total thyroidectomy. The rate of permanent hypoparathyroidism in quality registries are in the range of is 5-7 percent of patients undergoing surgery.

Patients operated on benign disease with total thyroidectomy, and who suffer from permanent hypoparathyroidism (defined as medication with active Vitamin D analogue therapy for more than 6 months, are at increased risk of renal insufficiency. They also have, for unclear reasons, an increased risk of suffering from malignancy, compared to patients without this complication. Patients with known ischemic heart disease before surgery also have an increased risk of suffering a new episode of cardiovascular disease. Finally, patients with permanent hypoparathyroidism have an increased risk of mortality compared to patients without this complication.

If, by using a technique for autofluorescence (Fluobeam® -LX), one can more accurately identify and avoid damage to the parathyroid glands during the surgical procedure, this would be of great importance for patients undergoing total thyroidectomy for thyroid disease.

Patients undergoing total thyroidectomy are randomized to the use of Fluobeam® -LX to detect the parathyroid glands through autofluorescence during thyroid surgery, or clinical evaluation only (control). Outcome is evaluated by parathyroid hormon (PTH) levels the first postoperative day and the need for medication with calcium and Vitamin D up to 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

Patients with thyroid disease planned for total thyroidectomy regardless of diagnosis

Exclusion Criteria:

* Previous thyroid surgery
* Previous parathyroid surgery
* Concurrent parathyroid surgery
* Renal insufficiency
* Pregnancy
* Breast feeding
* Allergy (contrast agent, iodine)
* Inability to understand study information
* Patient unable to participate in planned follow-up program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Postoperative level of Parathyroid hormone (PTH) | First postoperative day
  Low plasma parathyroid hormone (PTH) (below the normal reference range)

SECONDARY OUTCOMES:
Postoperative medication with Active vitamin D | At discharge (up to 7 days), at 1 month and at 6 months
  Medication with active Vitamin D; dihydrotachysterol (ATC A11CC02), alfacalcidol (ATC A11CC03), or calcitriol (ATC A11CC04) due to postoperative hypocalcaemia. Evaluated by standard questionaire in the database "Eurocrine" (yes/no)
Postoperative medication with oral calcium | At discharge (up to 7 days), at 1 month and at 6 months
  Medication with oral calcium; calcium carbonate (A12AA04), and calcium lactate gluconate (A12AA06) Evaluated by standard questionaire in the database "Eurocrine" (yes/no)
Identification of parathyroid glands | Intraoperatively
  Number of identified parathyroid glands
Autotransplantation of parathyroid tissue | Intraoperatively
  Number of autotransplanted parathyroid glands
Excised parathyroid glands | One week
  Number of excised parathyroid glands found on the specimen at histopathology
Time for operation | Intraoperatively
  Time for surgery (skin to skin) in minutes
Hospital stay | One week
  Hospital stay in days
Re-hospitalization due to hypocalcaemia | One month
  Any subsequent hospitalization within 30 days for hypocalcaemia-related symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Anders OJ Bergenfelz, PhD, Principal Investigator — Skane University Hospital
Locations (5):
- Rudolfstiftung, Vienna, Austria
- Haukeland University Hospital, Bergen, Norway
- Jagiellonian University Medical College, Krakow, Poland
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Skåne University Hospital, Department of Surgery, Lund, Lund

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in a publication. Individuals are de-identified
Supporting Information: Study Protocol
Time Frame: Starting 12 months after publication and for five years
Access Criteria: Researchers within the medical community The principal investigator or the Central Contact Backup will review requests.

REFERENCES:
- [Derived] Bergenfelz A, Barczynski M, Heie A, Muth A, Passler C, Schneider M, Wierzbicka P, Konturek A, Brauckhoff K, Elf AK, Dahlberg J, Hermann M. Impact of autofluorescence for detection of parathyroid glands during thyroidectomy on postoperative parathyroid hormone levels: parallel multicentre randomized clinical trial. Br J Surg. 2023 Nov 9;110(12):1824-1833. doi: 10.1093/bjs/znad278. PMID 37758507